CLINICAL TRIAL: NCT02136511
Title: An Expanded Access Protocol for Idelalisib in Combination With Rituximab for Relapsed, Previously Treated Subjects With Chronic Lymphocytic Leukemia
Brief Title: Expanded Access for Idelalisib in Combination With Rituximab in Chronic Lymphocytic Leukemia
Status: Approved for marketing | Type: Expanded Access
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-312-1325; 2013-005343-82 (EudraCT Number)
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; Rituximab

INTERVENTIONS:
Drug: Idelalisib — Idelalisib 150 mg tablet administered orally twice daily
  Other Names: GS-1101; CAL-101; Zydelig®
Drug: Rituximab — Rituximab administered intravenously starting at 375 mg/m^2 at Week 0 and continuing with a dose of 500 mg/m^2 at Weeks 2, 4, 6, 8, 12, 16, and 20.
  Other Names: Rituxan®

SUMMARY:
This study is to provide idelalisib (IDELA) to individuals with relapsed, previously treated chronic lymphocytic leukemia (CLL) who have limited treatment options and are not eligible for other Gilead-sponsored studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age with a diagnosis of B-cell CLL established according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria and documented within medical records
2. CLL that warrants treatment (consistent with accepted IWCLL criteria for initiation of therapy)
3. Prior treatment for CLL comprising any of the following:

   1. Prior treatment with ≥ 1 regimen containing a therapeutic anti-CD20 antibody or
   2. Prior treatment with ≥ 2 regimens containing ≥ 1 cytotoxic agent
4. CLL progression < 24 months since the completion of the last prior therapy for CLL
5. Appropriate for noncytotoxic-containing therapy based on the presence of any of the following factors:

   1. Grade ≥ 3 neutropenia or thrombocytopenia attributable to cumulative myelotoxicity from prior administration of cytotoxic agents (as documented by bone marrow biopsy obtained since last prior therapy), or
   2. Estimated creatinine clearance < 60 mL/min (as determined by the Cockcroft-Gault method), or
   3. A Cumulative Illness Rating Scale (CIRS) score of > 6
6. A negative serum pregnancy test for female subjects of childbearing potential
7. Male and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
8. Lactating females must agree to discontinue nursing before the study drug is administered.
9. Evidence of a personally signed informed consent

Exclusion Criteria:

1. Known hypersensitivity to the idelalisib, its metabolites, or formulation excipient(s)
2. Known histological transformation from CLL to an aggressive lymphoma (ie, Richter transformation)
3. Known myelodysplastic syndrome
4. Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of randomization
5. Ongoing drug-induced liver injury, chronic active hepatitis C (HCV), chronic active hepatitis B (HBV), alcoholic liver disease, nonalcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension
6. Ongoing drug-induced pneumonitis
7. Ongoing inflammatory bowel disease
8. History of anaphylaxis in association with previous administration of monoclonal antibodies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jahn, MD, Study Director — Gilead Sciences
Locations (8):
- United States (4):
  - University of California, San Diego - Moores Cancer Center, La Jolla, California
  - Georgetown University, Washington D.C., District of Columbia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
- St. James University Hospital, Dublin, Ireland
- Italy (2):
  - Ospedale San Raffaele, Milan
  - A.S.O. Molinette S. Giovanni Battista, Turin
- Hammersmith Hospital, London, United Kingdom